CLINICAL TRIAL: NCT04242498
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Bimekizumab in Study Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Study Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: BE HEARD II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS0004; 2019-002551-42 (EudraCT Number)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: Bimekizumab; UCB4940; HS; Hidradenitis Suppurativa; Acne inversa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bimekizumab dosing regimen 1 (Experimental): Subjects participating in the study will receive assigned bimekizumab dosing regimen 1 during the Treatment Period.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosing regimen 2 (Experimental): Subjects participating in the study will receive assigned bimekizumab dosing regimen 2 during the Treatment Period.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosing regimen 3 (Experimental): Subjects participating in the study will receive assigned bimekizumab dosing regimen 3 during the Treatment Period.
  Interventions: Drug: Bimekizumab
- Placebo Group (Placebo Comparator): Subjects randomized to this arm will receive placebo during the Initial Treatment Period and bimekizumab during the Maintenance Treatment Period.
  Interventions: Drug: Bimekizumab; Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: UCB4940
Other: Placebo — Subjects will receive placebo at pre-specified time-points during the Initial Treatment Period.
  Other Names: PBO
  Arms: Placebo Group

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of bimekizumab in study participants with moderate to severe hidradenitis suppurativa (HS)

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age, at the time of signing the informed consent. If a study participant is under the local age of consent and is at least 18 years of age, written informed consent will be obtained from both the study participant and the legal representative
* Study participants must have a diagnosis of Hidradenitis Suppurativa (HS) based on clinical history and physical examination for at least 6 months prior to the Baseline visit
* Study participant must have HS lesions present in at least 2 distinct anatomic areas (eg, left and right axilla), 1 of which must be at least Hurley Stage II or Hurley Stage III at both the Screening and Baseline visits
* Study participant must have moderate to severe HS defined as a total of ≥5 inflammatory lesions (ie, number of abscesses plus number of inflammatory nodules) at both the Screening and Baseline visits
* Study participant must have had an inadequate response to a course of a systemic antibiotic for treatment of HS as assessed by the Investigator through study participant interview and review of medical history
* A female study participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 20 weeks after the last dose of investigational medicinal product (IMP)

Exclusion Criteria:

* Draining tunnel count of >20 at the Baseline Visit
* Any other active skin disease or condition (eg, bacterial cellulitis, candida intertrigo, extensive condyloma) that may, in the opinion of the Investigator, interfere with the assessment of hidradenitis suppurativa (HS)
* Study participant has a diagnosis of sarcoidosis, systemic lupus erythematosus, or active inflammatory bowel disease (IBD)
* Primary immunosuppressive condition, including taking immunosuppressive therapy following an organ transplant, or has had a splenectomy
* Female who is breastfeeding, pregnant, or plans to become pregnant during the study or within 20 weeks following the final dose of investigational medicinal product (IMP)
* Active infection or history of certain infection(s)
* Active tuberculosis (TB) infection, latent TB infection, high risk of exposure to TB infection, current or history of nontuberculous mycobacterium (NTM) infection
* Concurrent malignancy. Study participants with a history of malignancy within the past 5 years prior to the Screening Visit are excluded, EXCEPT if the malignancy was a cutaneous squamous or basal cell carcinoma, or in situ cervical cancer that has been treated and is considered cured
* History of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease
* Known hypersensitivity to any components of bimekizumab or comparative drugs as stated in this protocol this protocol
* Concomitant and prior medication restrictions
* Myocardial infarction or stroke within the 6 months prior to the Screening Visit
* Study participant has the presence of active suicidal ideation, or positive suicide behavior using the "Screening" version of the electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
* Presence of moderately severe major depression or severe major depression
* Subject has a history of chronic alcohol or drug abuse within 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (91):
- United States (24):
  - Hs0004 50162, Fountain Valley, California
  - Hs0004 50196, Thousand Oaks, California
  - Hs0004 50199, Miami, Florida
  - Hs0004 50152, Orange Park, Florida
  - Hs0004 50144, Orlando, Florida
  - Hs0004 50184, Pembroke Pines, Florida
  - Hs0004 50193, Sandy Springs, Georgia
  - Hs0004 50223, Savannah, Georgia
  - Hs0004 50164, Skokie, Illinois
  - Hs0004 50234, Plainfield, Indiana
  - Hs0004 50178, Clarkston, Michigan
  - Hs0004 50105, St Louis, Missouri
  - Hs0004 50197, Henderson, Nevada
  - Hs0004 50159, Portsmouth, New Hampshire
  - Hs0004 50200, Verona, New Jersey
  - Hs0004 50237, Albuquerque, New Mexico
  - Hs0004 50211, Durham, North Carolina
  - Hs0004 50179, Winston-Salem, North Carolina
  - Hs0004 50145, Columbus, Ohio
  - Hs0004 50202, Fairborn, Ohio
  - Hs0004 50150, Philadelphia, Pennsylvania
  - Hs0004 50236, Greenville, South Carolina
  - Hs0004 50084, Johns Island, South Carolina
  - Hs0004 50148, Pflugerville, Texas
- Australia (3):
  - Hs0004 30018, Parkville
  - Hs0004 30014, St Leonards
  - Hs0004 30009, Westmead
- Bulgaria (6):
  - Hs0004 40313, Pleven
  - Hs0004 40284, Sofia
  - Hs0004 40311, Sofia
  - Hs0004 40314, Sofia
  - Hs0004 40315, Sofia
  - Hs0004 40353, Stara Zagora
- Canada (6):
  - Hs0004 50172, Cobourg
  - Hs0004 50135, Edmonton
  - Hs0004 50174, London
  - Hs0004 50189, St. John's
  - Hs0004 50134, Waterloo
  - Hs0004 50136, Winnipeg
- Czechia (2):
  - Hs0004 40063, Prague
  - Hs0004 40194, Prague
- France (9):
  - Hs0004 40245, Antony
  - Hs0004 40321, Auxerre
  - Hs0004 40129, Bordeaux
  - Hs0004 40320, La Rochelle
  - Hs0004 40247, Lyon
  - Hs0004 40130, Marseille
  - Hs0004 40404, Reims
  - Hs0004 40403, Saint-Etienne
  - Hs0004 40286, Toulouse
- Germany (8):
  - Hs0004 40289, Berlin
  - Hs0004 40326, Berlin
  - Hs0004 40322, Dessau
  - Hs0004 40356, Dresden
  - Hs0004 40287, Frankfurt am Main
  - Hs0004 40142, Hamburg
  - Hs0004 40328, Hanover
  - Hs0004 40250, Lübeck
- Hs0004 40254, Debrecen, Hungary
- Hs0004 40344, Dublin, Ireland
- Hs0004 20090, Afula, Israel
- Japan (13):
  - Hs0004 20196, Bunkyō City
  - Hs0004 20144, Fukuoka
  - Hs0004 20043, Itabashi-ku
  - Hs0004 20195, Kagoshima
  - Hs0004 20170, Kurume
  - Hs0004 20190, Kyoto
  - Hs0004 20033, Nagoya
  - Hs0004 20152, Nakagami-gun
  - Hs0004 20178, Nishinomiya
  - Hs0004 20153, Obihiro
  - Hs0004 20037, Osaka
  - Hs0004 20154, Sapporo
  - Hs0004 20171, Sendai
- Poland (6):
  - Hs0004 40347, Lodz
  - Hs0004 40293, Rzeszów
  - Hs0004 40335, Warsaw
  - Hs0004 40095, Wroclaw
  - Hs0004 40333, Wroclaw
  - Hs0004 40334, Wroclaw
- Spain (6):
  - Hs0004 40159, Barcelona
  - Hs0004 40267, Barcelona
  - Hs0004 40298, Granada
  - Hs0004 40268, Madrid
  - Hs0004 40297, Manises
  - Hs0004 40101, Sabadell
- United Kingdom (5):
  - Hs0004 40300, Cardiff
  - Hs0004 40339, Leeds
  - Hs0004 40113, London
  - Hs0004 40240, Newcastle upon Tyne
  - Hs0004 40338, Northampton

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Kirby JS, Thorlacius L, Lambert J, Ciaravino V, Rolleri R, Pansar I, Muller E, Pelligra CG, Ingram JR. Psychometric validation and interpretation thresholds of the Hidradenitis Suppurativa Quality of Life (HiSQOL(c)) questionnaire using pooled data from the phase III BE HEARD I & II trials of bimekizumab in hidradenitis suppurativa. Br J Dermatol. 2025 Jun 20;193(1):93-104. doi: 10.1093/bjd/ljaf067. PMID 40172122
- [Result] Ingram JR, Lambert J, Ciaravino V, Rolleri R, Pansar I, Peterson L, Pelligra CG, Thorlacius L. Hidradenitis Suppurativa Symptom Daily Diary (HSSDD) and Questionnaire (HSSQ): Psychometric Validation and Interpretation Threshold Derivation Using Phase 3 Study Data. Dermatol Ther (Heidelb). 2025 May;15(5):1093-1111. doi: 10.1007/s13555-025-01346-w. Epub 2025 Mar 28. PMID 40153232
- [Result] Shi VY, Ingram JR, Lev-Tov H, Schneider-Burrus S, Forman S, Porter ML, Hayama K, Thorlacius L, Lambert J, Vaux T, Lukowski B, Rolleri RL, Szepietowski JC. Bimekizumab Impact on Patient-Reported Outcomes in Patients with Moderate to Severe Hidradenitis Suppurativa: Pooled 48-Week Results from BE HEARD I&II. Dermatol Ther (Heidelb). 2025 Sep;15(9):2553-2570. doi: 10.1007/s13555-025-01465-4. Epub 2025 Jul 13. PMID 40652434
- [Result] Ingram JR, Fujita H, Gottlieb AB, Lev-Tov H, Prens E, Sayed CJ, Shi VY, Szepietowski JC, Takahashi K, Frew JW, Lambert J, Davis L, Oh T, Rolleri R, Saintmard MH, Orenstein LAV. Bimekizumab Pain Outcomes in Patients with Hidradenitis Suppurativa: Pooled 48-Week Results from BE HEARD I&II Phase 3 Randomized Clinical Trials. Pain Ther. 2025 Dec;14(6):1861-1878. doi: 10.1007/s40122-025-00779-7. Epub 2025 Oct 17. PMID 41107641
- [Derived] Kimball AB, Jemec GBE, Sayed CJ, Kirby JS, Prens E, Ingram JR, Garg A, Gottlieb AB, Szepietowski JC, Bechara FG, Giamarellos-Bourboulis EJ, Fujita H, Rolleri R, Joshi P, Dokhe P, Muller E, Peterson L, Madden C, Bari M, Zouboulis CC. Efficacy and safety of bimekizumab in patients with moderate-to-severe hidradenitis suppurativa (BE HEARD I and BE HEARD II): two 48-week, randomised, double-blind, placebo-controlled, multicentre phase 3 trials. Lancet. 2024 Jun 8;403(10443):2504-2519. doi: 10.1016/S0140-6736(24)00101-6. Epub 2024 May 22. PMID 38795716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2020 and concluded in September 2022.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS) and Maintenance Set (MS).
Groups:
- Placebo: Participants received placebo during the 16-weeks Initial Treatment Period.
- BKZ Dosing Regimen 1: Participants received Bimekizumab (BKZ) dosing regimen 1 subcutaneously (SC) during the 16-weeks Initial Treatment Period.
- BKZ Dosing Regimen 2: Participants received BKZ dosing regimen 2 SC during the 16-weeks Initial Treatment Period.
- Placebo/BKZ Dosing Regimen 2: After the 16-weeks Initial Treatment Period, participants initially randomized to placebo received BKZ dosing regimen 2 SC during the 32-weeks Maintenance Treatment Period (up to Week 48).
- BKZ Dosing Regimen 1/BKZ Dosing Regimen 1: After the 16-weeks Initial Treatment Period, participants initially randomized to BKZ dosing regimen 1 continued to receive BKZ dosing regimen 1 SC during the 32-weeks Maintenance Treatment Period (up to Week 48).
- BKZ Dosing Regimen 2/BKZ Dosing Regimen 1: After the 16-week Initial Treatment Period, participants initially randomized to BKZ dosing regimen 2 received BKZ dosing regimen 1 SC during the 32-weeks Maintenance Treatment Period (up to Week 48).
- BKZ Dosing Regimen 2/BKZ Dosing Regimen 2: After the 16-week Initial Treatment Period, participants initially randomized to BKZ dosing regimen 2 continued to receive BKZ dosing regimen 2 SC during the 32-weeks Maintenance Treatment Period (up to Week 48).
Period: Initial Treatment Period: Week 0-16
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2 | Placebo/BKZ Dosing Regimen 2 | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2
Started | 74 | 144 | 291 | 0 | 0 | 0 | 0
Completed | 69 | 133 | 262 | 0 | 0 | 0 | 0
Not Completed | 5 | 11 | 29 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 9 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Consent withdrawn by subject, not due to AE | 2 | 8 | 12 | 0 | 0 | 0 | 0
Not completed — Subject Moved Long Distance From Clinic (Abroad) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawn by investigator's decision | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized, not treated | 0 | 2 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Treatment Period: Week 16-48
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2 | Placebo/BKZ Dosing Regimen 2 | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2
Started | 0 | 0 | 0 | 69 | 133 | 130 | 131 (1 participant completed the 16-Week Initial Treatment Period but did not enter the Maintenance Treatment Period because of the below reason: consent withdrawn by subject (not due to adverse event).)
Completed | 0 | 0 | 0 | 61 | 109 | 107 | 110
Not Completed | 0 | 0 | 0 | 8 | 24 | 23 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 7 | 6 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 4 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 3 | 1 | 2
Not completed — Consent withdrawn by subject, not due to AE | 0 | 0 | 0 | 6 | 9 | 10 | 11
Not completed — Change In Address-Patient Not Wanting To Continue | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Visits Too Time-Consuming, Only SFU Will Be Done | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject Relocated | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the RS which consisted of all study participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2 | Total
Number analyzed (Participants) | 74 | 144 | 291 | 509
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 7 | 10 | 17
  Between 18 and 65 years | 70 | 135 | 277 | 482
  >=65 years | 4 | 2 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (13.2) | 35.2 (11.9) | 36.9 (12.3) | 36.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 77 | 150 | 258
  Male | 43 | 67 | 141 | 251
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 1 | 1
  Asian | 5 | 7 | 22 | 34
  Black | 5 | 13 | 22 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  White | 64 | 119 | 232 | 415
  Other/mixed | 0 | 4 | 12 | 16
  Missing | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 15 | 30
  Not Hispanic or Latino | 69 | 134 | 274 | 477
  Missing | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Response as Measured by Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) at Week 16
Description: HiSCR50 was defined as at least a 50 percent (%) reduction from Baseline in the total abscess and inflammatory nodule (AN) count, with no increase from Baseline in abscess or draining tunnel count. Intermittent missing data are imputed using multiple imputation with Markov Chain Monte Carlo (MCMC) method followed by monotone regression for monotone missing data. Lesion counts were imputed and then dichotomized to obtain the response status. Participants who experienced an intercurrent event were treated as nonresponders following the intercurrent event. An intercurrent event was defined as receipt of systemic antibiotic rescue medication or discontinuation of study treatment due to an adverse event (AE) or lack of efficacy. Percentages of participants shown do not account for model effects using the logistic regression model.
Time Frame: Week 16
Population: The RS consisted of all study participants randomized into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 144 | 291
percentage of participants | 32.2 [21.4 to 42.9] | 53.8 [45.4 to 62.1] | 52.0 [46.1 to 57.8]
Statistical Analysis 1: Comparison: Placebo vs BKZ Dosing Regimen 1; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.422, 97.5% CI 2-sided [1.221 to 4.804]
Statistical Analysis 2: Comparison: Placebo vs BKZ Dosing Regimen 2; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 2.287, 97.5% CI 2-sided [1.220 to 4.291]

2. Secondary Outcome: Percentage of Participants Achieving Clinical Response as Measured by Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) at Week 16
Description: HiSCR75 was defined as at least a 75% reduction from Baseline in the total AN count, with no increase from Baseline in abscess or draining tunnel count. Intermittent missing data were imputed using multiple imputation with MCMC method followed by monotone regression for monotone missing data. Lesion counts were imputed and then dichotomized to obtain the response status. Participants who experienced an intercurrent event were treated as nonresponders following the intercurrent event. An intercurrent event was defined as receipt of systemic antibiotic rescue medication or discontinuation of study treatment due to an AE or lack of efficacy. Percentages of participants shown do not account for model effects using the logistic regression model.
Time Frame: Week 16
Population: The RS consisted of all study participants randomized into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 144 | 291
percentage of participants | 15.6 [7.2 to 24.0] | 33.7 [25.7 to 41.7] | 35.7 [30.1 to 41.3]
Statistical Analysis 1: Comparison: Placebo vs BKZ Dosing Regimen 1; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.722, 97.5% CI 2-sided [1.182 to 6.267]
Statistical Analysis 2: Comparison: Placebo vs BKZ Dosing Regimen 2; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 3.007, 97.5% CI 2-sided [1.374 to 6.581]

3. Secondary Outcome: Percentage of Participants With Flare by Week 16
Description: Flare was defined as a greater than or equal to (>=) 25% increase in AN count with an absolute increase in AN count of >= 2 relative to Baseline. Intermittent missing data were imputed using multiple imputation with MCMC method followed by monotone regression for monotone missing data. Lesion counts were imputed and then dichotomized to obtain the response status. Participants who experienced an intercurrent event prior to experiencing a flare were treated as having experienced a flare at all flare assessments on and after the intercurrent event date. An intercurrent event was defined as receipt of systemic antibiotic rescue medication or discontinuation of study treatment due to an AE or lack of efficacy. Percentages of participants shown do not account for model effects using the logistic regression model.
Time Frame: From Baseline to Week 16
Population: The RS consisted of all study participants randomized into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 144 | 291
percentage of participants | 28.0 [17.6 to 38.4] | 23.6 [16.5 to 30.7] | 28.8 [23.5 to 34.1]
Statistical Analysis 1: Comparison: Placebo vs BKZ Dosing Regimen 1; Test type: Superiority; p = 0.497, Regression, Logistic; Odds Ratio (OR) = 0.798, 97.5% CI 2-sided [0.378 to 1.683]
Statistical Analysis 2: Comparison: Placebo vs BKZ Dosing Regimen 2; Test type: Superiority; p = 0.868, Regression, Logistic; Odds Ratio (OR) = 1.050, 97.5% CI 2-sided [0.541 to 2.041]

4. Secondary Outcome: Absolute Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: The DLQI is a patient-reported questionnaire designed for use in adult participants with skin diseases and Hidradenitis Suppurativa (HS). The DLQI is a skin disease-specific questionnaire aimed at the evaluation of how symptoms and treatment affect patients' health related quality of life (HRQoL), with a recall period of 7 days. This instrument asks participants 10 questions about symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The scoring of each answer for the DLQI is on a scale range of 0 (not at all) to 3 (very much). The DLQI total score was calculated by adding the score of each question. The maximum score is 30, and the minimum score is 0. The higher the score, the more quality of life is impaired. Participants who experienced an intercurrent event were treated as missing following the intercurrent event and imputed using the multiple imputation method for missing data.
Time Frame: Baseline, Week 16
Population: The RS consisted of all study participants randomized into the study. Mean values shown do not account for model effects using the analysis of covariance (ANCOVA) model. Intercurrent event defined as receipt of systemic antibiotic rescue medication or discontinuation of study treatment due to AE or lack of efficacy.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 144 | 291
score on a scale | -3.2 (0.6) | -4.7 (0.5) | -4.6 (0.3)
Statistical Analysis 1: Comparison: Placebo vs BKZ Dosing Regimen 1; Test type: Superiority; p < 0.001, ANCOVA — Nominal p-value only due to the testing hierarchy failing on the flare outcome; LS mean difference = -2.393, 97.5% CI 2-sided [-3.920 to -0.867]
Statistical Analysis 2: Comparison: Placebo vs BKZ Dosing Regimen 2; Test type: Superiority; p < 0.001, ANCOVA — Nominal p-value only due to the testing hierarchy failing on the flare outcome; LS mean difference = -2.309, 97.5% CI [-3.705 to -0.914]

5. Secondary Outcome: Absolute Change From Baseline in Worst Skin Pain Score at Week 16
Description: Absolute change from Baseline in worst Skin Pain score at Week 16 was assessed using the worst skin pain item in the Hidradenitis Suppurativa Symptom Daily Diary (HSSDD). Worst skin pain during the past 24 hours was assessed daily using an 11-point numeric rating scale (NRS) which ranges from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The worst skin pain score was derived from the weekly average of daily scores, defined as the sum of the scored item over the course of the study week divided by the number of days in which the item was completed, relative to each respective visit date. Intermittent missing data are imputed using multiple imputation with MCMC method followed by monotone regression for monotone missing data. Participants who experienced an intercurrent event were treated as missing following the intercurrent event and imputed using the multiple imputation method for missing data. Mean values shown do not account for model effects using the ANCOVA model.
Time Frame: Baseline, Week 16
Population: The RS consisted of all study participants randomized into the study. Intercurrent event defined as receipt of systemic antibiotic rescue medication or discontinuation of study treatment due to AE or lack of efficacy.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 144 | 291
score on a scale | -0.36 (0.30) | -1.44 (0.24) | -1.83 (0.17)
Statistical Analysis 1: Comparison: Placebo vs BKZ Dosing Regimen 1; Test type: Superiority; p = 0.010, ANCOVA — Nominal p-value only due to the testing hierarchy failing on the flare outcome; LS mean difference = -0.898, 97.5% CI 2-sided [-1.684 to -0.113]
Statistical Analysis 2: Comparison: Placebo vs BKZ Dosing Regimen 2; Test type: Superiority; p < 0.001, ANCOVA — Nominal p-value only due to the testing hierarchy failing on the flare outcome; LS mean difference = -1.265, 97.5% CI 2-sided [-1.978 to -0.552]

6. Secondary Outcome: Percentage of Participants Achieving Skin Pain Response at Week 16
Description: Skin pain response at Week 16, as assessed by "worst skin pain" item in HSSDD, was defined as an improvement in weekly worst skin pain score of at least 3 points versus Baseline. Worst skin pain during the past 24 hours was assessed daily using an 11-point numeric rating scale (NRS) which ranges from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). Worst skin pain score was derived from weekly average of daily scores (sum of scored item over study week/number of days in which item completed, relative to each respective visit). Intermittent missing data were imputed using multiple imputation with MCMC method followed by monotone regression for monotone missing data. Weekly pain scores were imputed and then dichotomized to obtain response status. Participants who experienced an intercurrent event were treated as non-responders following the intercurrent event. Percentages of participants shown do not account for model effects using logistic regression model.
Time Frame: Week 16
Population: The RS consisted of all study participants randomized into the study. Here, number of participants analyzed included RS with HSSDD worst skin pain score >=3 at Baseline. Intercurrent event defined as receipt of systemic antibiotic rescue medication or discontinuation of study treatment due to AE or lack of efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2
Number analyzed (Participants) | 49 | 108 | 209
percentage of participants | 10.9 [1.7 to 20.1] | 28.6 [19.5 to 37.8] | 31.8 [25.1 to 38.4]
Statistical Analysis 1: Comparison: Placebo vs BKZ Dosing Regimen 1; Test type: Superiority; p = 0.028, Regression, Logistic — Nominal p-value only due to the testing hierarchy failing on the flare outcome; Odds Ratio (OR) = 3.273, 97.5% CI 2-sided [0.974 to 10.997]
Statistical Analysis 2: Comparison: Placebo vs BKZ Dosing Regimen 2; Test type: Superiority; p = 0.010, Regression, Logistic — Nominal p-value only due to the testing hierarchy failing on the flare outcome; Odds Ratio (OR) = 3.756, 97.5% CI 2-sided [1.189 to 11.867]

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week Safety Follow-Up [SFU] period).
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 71)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP. The MS consisted of all study participants who received at least 1 dose (full or partial) of BKZ in the Maintenance Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2 | Placebo/BKZ Dosing Regimen 2 | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 142 | 290 | 69 | 133 | 130 | 131
percentage of participants | 56.8 | 51.4 | 64.5 | 71.0 | 72.2 | 77.7 | 77.1

8. Secondary Outcome: Percentage of Participants With Serious Treatment-emergent Adverse Events During the Study
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: Results in death; Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent disability/incapacity; Is a congenital anomaly/birth defect; Important medical events. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week SFU period).
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 71)
Population: The SS consisted of all study participants who received at least 1 dose (full or partial) of IMP. The MS consisted of all study participants who received at least 1 dose (full or partial) of BKZ in the Maintenance Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2 | Placebo/BKZ Dosing Regimen 2 | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 142 | 290 | 69 | 133 | 130 | 131
percentage of participants | 0 | 2.1 | 3.1 | 2.9 | 3.0 | 2.3 | 3.1

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal From the Study
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week SFU period). TEAEs leading to discontinuation of the study are reported.
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 71)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2 | Placebo/BKZ Dosing Regimen 2 | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2
Number analyzed (Participants) | 74 | 142 | 290 | 69 | 133 | 130 | 131
percentage of participants | 0 | 2.1 | 4.1 | 0 | 4.5 | 3.1 | 1.5

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 71)
Description: Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week SFU period). TEAEs were analyzed and reported for Initial Treatment Period (SS) and Maintenance Treatment Period (MS) separately.
Arm/Group | Placebo | BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2 | Placebo/BKZ Dosing Regimen 2 | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/142 | 0/290 | 0/69 | 0/133 | 0/130 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/74 | 3/142 | 9/290 | 2/69 | 4/133 | 3/130 | 4/131
Other Adverse Events (participants affected / at risk) | 18/74 | 40/142 | 101/290 | 26/69 | 49/133 | 57/130 | 64/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=74) | BKZ Dosing Regimen 1 (N=142) | BKZ Dosing Regimen 2 (N=290) | Placebo/BKZ Dosing Regimen 2 (N=69) | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 (N=133) | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 (N=130) | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2 (N=131)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=74) | BKZ Dosing Regimen 1 (N=142) | BKZ Dosing Regimen 2 (N=290) | Placebo/BKZ Dosing Regimen 2 (N=69) | BKZ Dosing Regimen 1/BKZ Dosing Regimen 1 (N=133) | BKZ Dosing Regimen 2/BKZ Dosing Regimen 1 (N=130) | BKZ Dosing Regimen 2/BKZ Dosing Regimen 2 (N=131)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 5 (6) | 18 (21) | 2 (3) | 6 (8) | 4 (5) | 3 (3)
Oral candidiasis (Infections and infestations) | 0 (0) | 5 (5) | 24 (26) | 3 (3) | 11 (13) | 16 (18) | 14 (17)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 8 (8) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 3 (3)
Headache (Nervous system disorders) | 7 (9) | 7 (9) | 18 (21) | 3 (3) | 7 (10) | 4 (5) | 7 (7)
Hidradenitis (Skin and subcutaneous tissue disorders) | 5 (6) | 13 (15) | 23 (27) | 7 (11) | 16 (19) | 24 (33) | 15 (15)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 11 (11) | 2 (2) | 6 (6) | 8 (9) | 11 (15)
Folliculitis (Infections and infestations) | 0 (0) | 5 (5) | 8 (9) | 2 (2) | 5 (8) | 6 (6) | 9 (11)
Corona virus infection (Infections and infestations) | 0 (0) | 3 (3) | 11 (11) | 4 (4) | 2 (2) | 7 (7) | 8 (8)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 5 (6) | 4 (4) | 7 (7) | 5 (6) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 9 (10) | 4 (4) | 5 (6) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT04242498/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT04242498/SAP_001.pdf